CLINICAL TRIAL: NCT01781182
Title: Infant Antibiotic Resistance and Implications for Therapeutic Decision-making
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Sharon Meropol, MD, PhD, Assistant Professor of Pediatrics and Epidemiology and Biostatistics9, University Hospitals Cleveland Medical Center
Other Study IDs: 1K23AI097284-01A1 (NIH); 1K23AI097284-01A1 (NIH)
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Bacterial Infections and Mycoses
MeSH Terms: conditions — Bacterial Infections and Mycoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — specific cultured antibiotic resistant organisms of interest Stool specimens Stool DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
Escalating resistance to antibiotics among disease-causing community bacteria increasingly threatens our ability to treat patients' infections. At the level of the physician-patient encounter, incentives at the patient level often take priority to society; this is often the case with antibiotic prescribing. Each patient level antibiotic treatment decision is based on how we value potential outcomes, including short-term benefits and risks and longer-term risks, including those related to future bacterial resistance to antibiotics. Unfortunately, antibiotics are often prescribed for illnesses unlikely to have a bacterial etiology; even a very small likelihood of benefit seems to outweigh an increased risk of future antibiotic resistance. While short-term effects of antibiotics on colonization with resistant bacteria have been demonstrated, the overall implications of each treatment for future individual, family and societal-level resistance remain difficult to quantify, and are often steeply discounted or ignored during decision-making. Knowledge regarding the longer-term effects of personal and household antibiotic use could better quantify these future resistance-related risks, and help guide antibiotic decision-making for physicians and patients.

Infants are born with sterile nasopharyngeal and gastrointestinal tracts and yet, during the 1st year of life, become important reservoirs of resistant organisms; this creates an opportunity to study colonization and resistance starting from a microbiological tabula rasa. In this proposal, we will use an observational cohort to following newborns' antibiotic exposure and longitudinal colonization with specific bacterial pathogens and related antibiotic resistance in the 1st year of life. Our hypothesis is that during the 1st year of life, infants with personal and household antibiotic exposure will have greater colonization with resistan organisms than infants without antibiotic exposure. This project will help us understand the development of bacteria that are resistant to antibiotics within the community, and help to inform judicious decision-making regarding antibiotic prescribing.

ELIGIBILITY:
Inclusion Criteria:

* Infant in regular nursery at University Hospitals CWRU
* Mother has legal custody
* Mother is >=18 years old
* Mother's and baby's physicians have granted permission for possible enrollment
* Mother speaks, reads and understands the English language

Exclusion Criteria:

* Does not fit inclusion criteria

Max Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborn infants from the well baby nursery, followed during their first year of life
Sampling Method: Non-Probability Sample
Enrollment: 352 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Colonization with resistant organism of interest | First 12 months of life

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States